CLINICAL TRIAL: NCT03767985
Title: A Randomised Clinical Trial Objectively Comparing the Effect of Patching Therapy With Video Gaming for Amblyopia
Brief Title: Patching or Gaming as Amblyopia Treatment?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Lijf & Leven (Unknown); ODAS Stichting (Unknown); Uitzicht (Unknown); University of Applied Sciences Utrecht (Other)
Responsible Party: Principal Investigator, Sjoukje Elizabeth Loudon, MD, PhD, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MEC-2016-439
Record Dates: First submitted 2018-12-06; First posted 2018-12-07 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Intervention Model Description: Participants are randomized to either the standard patching therapy or the dichoptic video game therapy.
Who Masked: Care Provider
Masking Description: The research orthoptist that does the orthoptic examinations is masked to the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Occlusion therapy (Active Comparator): Participants are prescribed 2 hours of occlusion therapy per day, 7 days a week.
  Interventions: Other: Occlusion therapy
- Dichoptic video game therapy (Experimental): Participants receive dichoptic video game therapy: 1 hour per week at the out-patient clinic under direct supervision.
  Interventions: Other: Dichoptic video game therapy

INTERVENTIONS:
Other: Dichoptic video game therapy — Dichoptic video gaming for 1 hour per week, viewed through the Oculus Rift.
  Arms: Dichoptic video game therapy
Other: Occlusion therapy — Occlusion therapy for 2 hours per day, 7 days a week
  Arms: Occlusion therapy

SUMMARY:
Amblyopia affects 3% of the children and is caused by strabismus, anisometropia or both. Standard treatment is glasses and patching therapy. From North-America, behavioural training, i.e. dichoptic training, perceptual learning and video gaming, has become increasingly popular to improve visual acuity not only in children but also in adults. In this study we aim to compare the standard occlusion therapy with dichoptic video gaming.

DETAILED DESCRIPTION:
Amblyopia affects 3% of the children and is caused by strabismus, anisometropia or both. The standard treatment is glasses and patching therapy. From North-America, behavioural training, i.e. dichoptic training, perceptual learning and video gaming, has become increasingly popular. The rationale behind these games is by using dichoptic stimulation, with the contrast of the stimuli presented to the good eye reduced to match the appearance of the same stimuli when shown to the amblyopic eye, suppression can be alleviated. The many studies now conducted, demonstrate improvement in visual acuity with the games, the effect however is limited, but the rate of improvement is higher. In these studies, prescribed patching-time was compared to realised game-time. We have demonstrated in multiple studies that electronically measured compliance is low: on average only 50%.

In this study we aim to compare the effect of patching therapy, using the ODM to objectively measure compliance, with the effect of a novel dichoptic action video game in children as well as in adults. In addition, the adult participants will undergo fMRI scans to document any changes in the visual cortex before and after either therapy.

ELIGIBILITY:
Inclusion Criteria:

* Amblyopia; an interocular difference in visual acuity of at least 2 logMAR lines.

Exclusion Criteria:

* A non-comitant or large angle constant strabismus >30Prism Dioptres, a neurological disorder, nystagmus, other eye disorders and diminished acuity due to medication, brain damage or trauma.

Ages: 4 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 124 (Estimated)
Dates: Start 2017-12-18 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity improvement | 24 weeks
  Visual Acuity improvement (logMAR units/time period) in children with amblyopia treated with patching therapy vs dichoptic video gaming

CONTACTS AND LOCATIONS:
Overall Officials: Johannes R Vingerling, MD, PhD, Study Director — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tan ET, Kadhum A, Telleman MA, Treur A, Bruijning J, Loudon SE. How do parents experience patching or dichoptic action video gaming as amblyopia treatment? A qualitative study exploring treatment preferences and information needs to facilitate decision-making. Ophthalmic Physiol Opt. 2023 Jul;43(4):649-659. doi: 10.1111/opo.13132. Epub 2023 Apr 3. PMID 37010918